CLINICAL TRIAL: NCT06487494
Title: Is 2-Octyl Cyanoacrylate (2-OCA) With Four Interrupted Sutures Non-inferior to Continuous Suturing as a Wound Closure Technique in Adult Male Circumcision: A Randomized Controlled Pilot Study
Brief Title: Evaluating the Efficacy of 2-Octyl Cyanoacrylate (2-OCA) With Four Interrupted Sutures in Adult Male Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Premal Patel, MD, Assistant Professor, Department of Surgery. Director, Undergraduate Urologic Medical Education, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS26545
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2024-07

CONDITIONS: Phimosis; Paraphimosis
MeSH Terms: conditions — Phimosis; Paraphimosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2-octyl cyanoacrylate glue with four interrupted sutures (Experimental): In this arm the provider will use 2-octyl cyanoacrylate glue with four interrupted sutures for wound closing following circumcision.
  Interventions: Procedure: Circumcision wound closure using 2-octyl cyanoacrylate glue with four interrupted sutures
- Continuous suture (Active Comparator): In this arm the provider will use continuous suturing for wound closing following circumcision.
  Interventions: Procedure: Circumcision wound closure using continuous sutuing

INTERVENTIONS:
Procedure: Circumcision wound closure using 2-octyl cyanoacrylate glue with four interrupted sutures — 2-octyl cyanoacrylate glue is a wound closure adhesive which will be used with four interrupted sutures following circumcision for wound closure.
  Arms: 2-octyl cyanoacrylate glue with four interrupted sutures
Procedure: Circumcision wound closure using continuous sutuing — Continuous suturing is the standard following circumcision for wound closure.
  Arms: Continuous suture

SUMMARY:
This study aims to determine whether cyanoacrylate glue is a non-inferior alternative to continuous suturing for wound closure following adult circumcision. The primary objective of this study is to evaluate and compare operative time, pain, cosmesis, complications and patient satisfaction associated with the use of cyanoacrylate glue versus standard suturing for wound closure. To the best of our knowledge, this will be one of the first studies to investigate the use of cyanoacrylate glue for wound closure following adult circumcision. The findings from this study could provide valuable insights into the potential benefits of using cyanoacrylate glue as a non-inferior alternative to continuous suturing for wound closure. Additionally, this study may also inform clinical practice guidelines on the most effective techniques for wound closure following adult circumcision.

DETAILED DESCRIPTION:
This non-blinded, randomized controlled pilot study is to be conducted at the Men's Health Clinic in Winnipeg, Manitoba. All eligible patients undergoing circumcision will be invited to participate in the study. They will be randomly assigned in a 1:1 ratio using a computer-generated random list. Patients will be randomized to 2-Octyl cyanoacrylate (2-OCA) with four interrupted sutures vs. standard suturing alone. In the post-operative recovery area, patients will be asked to complete a VAS questionnaire. Patients will then be brought in for their routine visit 6 weeks post-op. During the visit, closure of the wound as well as any potential complications will be assessed by a research team member. At that time, a questionnaire will be administered to study participants to assess variables such as post-procedure pain as well as their satisfaction with the recovery process and cosmesis post-circumcision. Cosmesis and complications will also be assessed 12 weeks post-op.

ELIGIBILITY:
Inclusion Criteria:

* Patients >16 years of age undergoing circumcision will be included.

Exclusion Criteria:

* Patients <16 years of age who did not provide consent to be randomized.

Ages: 16 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Cosmesis | 6 and 12 weeks post-operation
  A cosmetic appearance satisfaction questionnaire will be administered at weeks 6 and 12 post-operation.
Post-operative Pain | Immediately post-operation and 6 weeks post-operation
  Using a visual analogue pain scale [range 0-10; 0 = no pain, 10 = maximal pain], pain will be assessed as reported by the patient to determine their pain.
Complication Rate | 6 and 12 weeks post-operation
  Measuring and recording any adverse events post procedure such as surgical site infection, bleeding, hematoma, diffuse swelling, and increased sensitivity amidst intercourse.
Intra-Operative Time | During the operation
  Intra-operative time will be measured starting when the physician makes the first incision and ends when sutures are finished.

CONTACTS AND LOCATIONS:
Locations (1):
- Men's Health Clinic Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No